CLINICAL TRIAL: NCT06825325
Title: Effect of Music on Pain Relief, Anxiety Reduction, and Feelings of Safety in Patients Undergoing Wound Debridement
Brief Title: Effect of Music During Wound Debridement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Serpil Uyar, Asst. Prof., Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024/505
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Debridement
Keywords: Debridement; Music; Pain; Anxiety; Sense of Safety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in the control group will not be allowed to listen to music. These patients will receive standard health care in the Diabetic Foot and Wound Care Clinic.
- Intervention Group- Listening to Sufi Music (Experimental): Patients in this group will listen to Sufi music for 15 minutes before the wound debridement in addition to standard health care in the Diabetic Foot and Wound Care Clinic. Music will be played to the patients with the help of Mp3 player and headphones. Disposable headphone covers will be used for the headphones and the covers will be changed for each patient.
  Interventions: Other: Music Listening

INTERVENTIONS:
Other: Music Listening — Selection of Sufi music will be played to the patients before the wound debridement.
  Arms: Intervention Group- Listening to Sufi Music

SUMMARY:
This randomized controlled intervention study aims to investigate the effect of music played before the debridement on patients' anxiety, pain, and sense of safety.

The study will be carried out with two groups: The control and the intervention groups with 100 participants for each group. While the control group participants will receive standard care, the intervention group participants will listen to selection of Sufi music before the debridement in addition to standard care.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM) is a chronic metabolic disease characterized by hyperglycemia caused by impaired insulin release, insulin action or both of these factors. The International Diabetes Federation Diabetes Atlas reports present global epidemiologic and diabetes-related impact data. According to the global findings of IDF 2021, 537 million adults (aged 20-79) are living with diabetes, representing 1 in 10 people. This number is projected to increase to 643 million by 2030 and 783 million by 2045.

Diabetes, which is becoming more and more common day by day, has many complications. One of the most important and most common chronic complications is "diabetic foot". The World Health Organization (WHO) recommends grouping all foot complications of diabetes, including the ankle, under the name "diabetic foot". The risk of a person with diabetes being admitted to hospital with a foot wound at any point in their life is approximately 35%. Foot ulcers in diabetics are recognized as an important health problem worldwide. Although diabetic foot ulcers are a preventable complication with preventive measures, when they develop, the treatment process is difficult and costly, and it is a major problem that causes limb loss and increased morbidity and mortality.

Debridement, which is a treatment method in diabetic foot wounds, basically contributes to rapid wound healing by turning the chronic wound into an acute wound. Debridement stimulates the tissue and removes the biofilm layer, foreign body and foreign material from the wound. In addition, debridement allows detailed evaluation of the wound and, if necessary, appropriate wound culture. The types of debridement in the literature are surgical, sharp, mechanical, biological, enzymatic and autolytic debridement. Sharp debridement is the removal of all unwanted components from the wound area with a scalpel, scissors or similar cutting instruments. It is an effective method that can be applied at the patient's bedside or in outpatient clinics, does not take time and can be defined as minor surgical intervention.

Debridement should be performed by a clinician specialized in the wound. One of the common problems encountered during sharp debridement in patients with diabetic foot is pain. Pain is included in our nursing diagnoses and can be managed by nurses. Unresolved pain in wound patients significantly affects wound healing, patient compliance with treatment and quality of life. Although sharp debridement is performed at the patient's bedside or in the outpatient clinic and does not require hospitalization, it causes the patient to experience anxiety. In addition, if the pain and anxiety experienced cannot be controlled, it causes a delay in the healing process.

In healthcare, all procedures are designed to restore patients' health, but the essential need for a sense of safety is often overlooked. It is the responsibility of healthcare professionals to foster a sense of safety in patients. When patients feel safety, it leads to numerous positive outcomes, such as improved healthcare delivery, increased patient satisfaction, and enhanced trust in the treatment process.

Traditional and complementary treatments refer to methods that support health needs outside of modern medicine, shaped by various cultures, religions, and beliefs. These treatments are classified into five categories, encompassing over 200 different approaches. One category, body-mind interventions, includes practices such as music, painting, dance, praying, and hypnosis. Music, as part of body-mind interventions, is processed by the temporal lobe and auditory center in the brain. It triggers physiological responses through the limbic system, which can reduce pain intensity by boosting endorphin release.

The literature review revealed a gap in research regarding the impact of music on patients' sense of safety. While numerous studies have explored music's effects on pain management, anxiety, and various diseases, no studies were found specifically examining the role of music in promoting a sense of safety. In Chittoria's study, patients listened to music during dressing and wound debridement as part of an additional intervention, for 10 minutes, three times a day. The results showed a slight reduction in blood pressure and pulse rate when debridement and dressing were performed with music. However, no studies were identified that assessed the combined effects of music on pain, anxiety, and the sense of safety in patients undergoing wound debridement. Understanding these interactions could offer healthcare professionals valuable insights, allowing them to manage pain, anxiety, and security more effectively and consciously.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or above,
* Visiting the hospital due to diabetic foot,
* Requiring wound debridement,
* Having wound debridement at least once before,
* Without hearing/speech impairment,
* Without a diagnosis of psychiatric disorders,
* Without any professional training in music,
* and volunteered to participate.

Exclusion Criteria:

* Patients under 18 years of age,
* Visiting the hospital for other wound causes,
* Having debridement before and after toe amputation,
* Having wound debridement for the first time
* With hearing/speech impairment,
* With a diagnosis of psychiatric disorders,
* With any kind of professional training in music,
* and not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-26 (Estimated); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale-Pain (NRS-P) | 15 minutes before the procedure and 5 minutes after the procedure
  The Numerical Rating Scale-Pain (NRS-P) is a one-dimensional tool that uses 11 numbers, ranging from 0 to 10, to assess pain intensity. The patient selects the number that most accurately reflects the severity of their pain, with 0 representing "no pain" and 10 indicating "the worst (unbearable) pain". The NRS-P is widely recognized as an effective method for measuring pain intensity, and it is generally considered more valid and reliable than other pain assessment scales.
Numerical Rating Scale-Anxiety (NRS-A) | 15 minutes before the procedure and 5 minutes after the procedure
  The Numerical Rating Scale-Anxiety (NRS-A) has been widely used in research to assess anxiety levels, with its reliability and validity well-established. This scale, which ranges from 0 to 10, measures anxiety from "No Stress" (0) to "Very Bad Stress" (10). A higher score indicates a greater level of anxiety. The scale categorizes raw anxiety scores as follows: 0-no anxiety, 1-3-slightly anxious, 4-6-moderately anxious, 7-9-very or extremely anxious, and 10-the worst imaginable or extremely anxious.

SECONDARY OUTCOMES:
Safety Feeling Scale | 15 minutes before the procedure and 5 minutes after the procedure
  Safety Feeling Scale, developed by Dabaghi et al. in 2023, is designed to assess the sense of security among hospitalized adult patients. It includes four sub-dimensions: effective care (5 items), trust in the healthcare team (3 items), emotional enrichment (2 items), and hygienic facilities (2 items), totaling 12 items. The scale uses a five-point Likert scale for responses:
  * Strongly disagree
  * Disagree
  * Undecided
  * Agree
  * Strongly agree Raw scale scores range from 12 to 60, with higher scores indicating a stronger sense of safety experienced by the patient in the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Serpil UYAR, Asst. Prof., Principal Investigator — Afyonkarahisar Health Sciences University